CLINICAL TRIAL: NCT01708863
Title: A Prospective Study of Patients With Hypoplastic Left Heart Syndrome (HLHS) Following Stage II Surgical Palliation
Status: Completed | Type: Observational
Sponsor: Timothy J Nelson, MD, PhD (Other)
Collaborators: University of Oklahoma (Other); Children's Hospital of Philadelphia (Other); Mayo Clinic (Other)
Responsible Party: Sponsor-Investigator, Timothy J Nelson, MD, PhD, Program Director, ReGen Theranostics, Inc.
Organization: ReGen Theranostics, Inc. (Other)
Other Study IDs: 12-002887
Record Dates: First submitted 2012-10-15; First posted 2012-10-17 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Hypoplastic Left Heart Syndrome
Keywords: Hypoplastic Left Heart Syndrome; Stage II palliative surgery; Glenn procedure; Congenital heart defect; Congenital heart disease; Underdeveloped left ventricle
MeSH Terms: conditions — Hypoplastic Left Heart Syndrome; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children with Hypoplastic Left Heart Syndrome (HLHS): HLHS patients requiring Stage II Glenn surgery

SUMMARY:
Hypoplastic left heart syndrome (HLHS) is a severe form of congenital heart disease that consists of multiple obstructions to flow through the left heart and aorta, as well as hypoplasia of the left ventricle. Most patients require a three-stage surgical protocol starting within days of birth. Stage I of this process is the Norwood reconstruction (within the first few days of life), Stage II (usually required within 3-8 months) involves creation of a direct connection between the patient's superior vena cava and the pulmonary arterial confluence (bidirectional Glenn anastomosis), and the last stage is creation of a Fontan circulation (typically within the first 2-4 years). This "single ventricle" approach requires the right ventricle to perform as the only circulatory pump for the entire body.

Our long-term goal is to develop regenerative strategies to strengthen and augment the right ventricular muscle of the single-ventricle heart following surgical palliation in HLHS patients. To determine the safety and feasibility of a cell-based therapeutic intervention at the Stage II surgery, we aim to document the natural history of post-surgical care in HLHS patients having undergone standard of care with protocol specific follow-up over the course of a 6-month period.

This prospective study will document the natural history in patients with HLHS after planned Stage II surgical palliation with a focus on cardiovascular parameters within 6 months following surgery in 10 patients.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with HLHS having undergone Stage I surgical palliation and undergoing planned Stage II palliative Glenn surgery.
* Individuals up to 18 months of age are eligible if written informed consent can be obtained from both parents and/or legal guardians, unless one parent is not reasonably available.

Exclusion Criteria:

* Severe chronic diseases, extensive extra-cardiac syndromic features, or history of cancer

The following complications of congenital heart disease:

* Any condition requiring urgent, or unplanned procedure within 15 days prior to Stage II surgical repair.
* Severe pulmonary hypertension (reported in the medical record as >70% systemic pressure).
* Other clinical concerns as documented by a site investigator that would predict (more likely to happen than not to happen) a risk of severe complications or very poor outcome during or after Stage II surgical repair.

Ages: 0 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with HLHS up to 18 months of age requiring a planned Stage II bi-directional Glenn surgery
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2020-05 (Actual); Study Completion 2020-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Nelson, MD, PhD, Study Director — Mayo Clinic; Muhammad Y Qureshi, MBBS, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic, Rochester, Minnesota
  - Oklahoma University Children's Hospital, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials